CLINICAL TRIAL: NCT04894071
Title: A Phase 1, Randomized, Double-Masked, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral QA102 in Healthy Young and Older Adult Subjects
Brief Title: QA102 Phase 1 Study in Healthy Young and Older Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Smilebiotek Zhuhai Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QA102-CS101
Record Dates: First submitted 2021-05-06; First posted 2021-05-20 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QA102 group (Experimental)
  Interventions: Drug: QA102
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QA102 — Intervention of Part 1: 6 dose levels (50mg, 100mg, 200mg, 400mg, 800mg, 1600mg of QA102 capsules), oral administration, single dose.
  Intervention of Part 2: 2 dose levels (the dose levels, dosing frequency and dosing duration will be decided on the basis of data from Part 1 of the study), oral administration.
  Intervention of Part 3: 1 dose level (the dose levels, dosing frequency and dosing duration will be decided on the basis of data from Part 2 of the study), oral administration.
  Arms: QA102 group
Drug: Placebo — Intervention of Part 1: 6 dose levels (50mg, 100mg, 200mg, 400mg, 800mg, 1600mg of Placebo capsules), oral administration, single dose.
  Intervention of Part 2: 2 dose levels (the dose levels, dosing frequency and dosing duration will be decided on the basis of data from Part 1 of the study), oral administration.
  Intervention of Part 3: 1 dose level (the dose levels, dosing frequency and dosing duration will be decided on the basis of data from Part 2 of the study), oral administration.
  Arms: Placebo group

SUMMARY:
This will be a double masked, randomized, placebo controlled, single and multiple oral dose study conducted in 3 parts. The safety and tolerability of single and multiple ascending oral doses of QA102 in healthy young and older adult subjects will be evaluated. The study will also characterize the pharmacokinetic (PK) profile of QA102 in plasma and urine after single and multiple oral doses of QA102. Besides, the metabolite profile of QA102 will also be characterized.

Part 1 will comprise a single dose, sequential cohort design. Part 2 will comprise a multiple dose, sequential cohort study. Part 3 will comprise a multiple dose, single cohort study in older subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index between 18.0 and 32.0 kg/m2, inclusive.
2. In good health, determined by no clinically significant findings from medical history, physical examination, visual acuity testing, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations at screening and check in as assessed by the investigator or designee.
3. Females of nonchildbearing potential defined as permanently sterile or postmenopausal. Males will agree to use contraception.
4. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
5. Young (between 18 and 59 years of age, for Part 1 and 2) or Older (between 60 and 75 years of age, for Part 3) males or females of nonchildbearing potential, of any race, inclusive, at screening.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
3. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
4. Active or recent (within 30 days of screening) infection or history of recurrent chronic infections with underlying condition that may predispose one to infections. Viral infections with symptoms resolved will be allowed up to 14 days prior to check-in.
5. History of malignancy of any type, other than surgically excised non-melanomatous skin cancers or in situ cervical cancer within 5 years before check-in.
6. Female subjects (surgically sterile females only) with a positive pregnancy test at screening or check in or who are lactating.
7. History of alcoholism or drug/chemical abuse within 2 years prior to check in.
8. Positive urine drug or alcohol results at screening or check in.
9. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives (whichever is longer) prior to dosing.
10. Consumption of alcohol from 48 hours prior to check-in.
11. Administration of any vaccine, including a Coronavirus Disease 2019 vaccine, within the past 30 days prior to dosing.
12. Subjects who, in the opinion of the investigator (or designee), should not participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events | Up to 7 days after dosing
  To evaluate the safety and tolerability of single and multiple ascending oral doses of QA102 in healthy young adult and elderly subjects.

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) from time zero to 12 hours postdose [AUC0-12] | up to 12 hours postdose
Maximum observed plasma concentration [Cmax] | Up to 48 hours postdose
time of the maximum observed plasma concentration [tmax] | up to 48 hours postdose

OTHER OUTCOMES:
renal clearance (CLR ) | up to 24 hours postdose
Metabolite characterization of QA102 | Within 24 hours after last dose
  To characterize metabolites of QA102 in plasma samples after multiple oral doses of QA102 in healthy adult subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No